CLINICAL TRIAL: NCT00719329
Title: Bacterial Colonization of the Neonatal Umbilical Cord and Impact of 4.0% Chlorhexidine Cleansing on the Bacteriological Profile of the Umbilical Cord of Newborns in Sylhet District, Bangladesh
Brief Title: Impact of Chlorhexidine Cleansing on Bacteria Colonizing the Umbilical Cord of Infants in Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Dhaka Shishu Hospital (Other); Shimantik, Bangladesh (Unknown); Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Luke C. Mullany, Associate Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: THRASHER-02827-0
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Results first posted 2012-04-20 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-03

CONDITIONS: Infection
Keywords: chlorhexidine; umbilical cord
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Chlorhexidine cleansing of the cord for seven days
  Interventions: Drug: Chlorhexidine 4.0%
- B (Experimental): Chlorhexidine cleansing of the cord for 1 day
  Interventions: Drug: Chlorhexidine 4.0%
- C (Placebo Comparator): Dry cord care, as recommended by WHO
  Interventions: Behavioral: Dry Cord Care

INTERVENTIONS:
Drug: Chlorhexidine 4.0% — Solution (4.0%, 7.1% CHX-D)
  Arms: A; B
Behavioral: Dry Cord Care — Educational messages regarding clean cord care
  Arms: C

SUMMARY:
Background: In developing countries, many babies are born at home and the umbilical cord commonly becomes infected during the first week after birth, and can be deadly. Cleansing of the cord with a low-cost antiseptic like chlorhexidine may reduce the risk of these infections. Little is known, however, about the frequency of chlorhexidine cleansing needed to impact upon the overall presence of bacteria on the stump, or regarding the changes in bacteria during the first week of life when most cord infections occur.

Objectives: We will describe the profile of bacteria colonizing the umbilical cord stump of infants in rural Bangladesh and examine the role of topical chlorhexidine in altering colonization and progress of infection. We will compare the overall and bacteria-specific rate of colonization of the cord stump between infants receiving chlorhexidine cleansing of their cord through the first day or first week of life. We will also quantify the relationship between colonization of the cord stump with specific pathogens and the presence and severity of signs of umbilical cord infection (pus, redness, swelling) among these newborns.

Potential Impact: More information is needed on the impact of single versus repeated applications of chlorhexidine to the cord stump, as the number of cleansing may substantially influence the feasibility of widespread scale-up in many populations. The data generated from this proposed study will guide the most appropriate design of this simple intervention and will help inform specific treatment protocols for effective management of infants with signs of umbilical cord infections.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in parent chlorhexidine cleansing trial

Exclusion Criteria:

* Not enrolled in parent trial
* First visited after 48 hours of life

Max Age: 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1931 (Actual)
Dates: Start 2008-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luke C Mullany, PhD, Study Director — Johns Hopkins Bloomberg School of Public Health
Locations (3):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States
- Bangladesh (2):
  - Projahnmo, Sylhet, Sylhet Division
  - Dhaka Shishu Hospital, Dhaka

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All babies recruited between September 2008 and September 2009
Pre-assignment Details: Babies were allocated based on their cluster allocation (i.e. location of birth) in the parent trial
Groups:
- CHX Cleansing - 7 Days: Chlorhexidine cleansing of the cord for seven days
- CHX Cleansing - 1 Day: Chlorhexidine cleansing of the cord for 1 day
- Dry Cord Care: Dry cord care, as recommended by WHO
Period: Overall Study
Arm/Group | CHX Cleansing - 7 Days | CHX Cleansing - 1 Day | Dry Cord Care
Started | 705 | 571 | 647
Day 1 Swab | 705 | 569 | 646
Day 3 Swab | 614 | 501 | 578
Day 7 Swab | 593 | 467 | 561
Completed | 705 | 569 | 646
Not Completed | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CHX Cleansing - 7 Days | CHX Cleansing - 1 Day | Dry Cord Care | Total
Number analyzed (Participants) | 705 | 571 | 647 | 1923
Age, Customized [Number; unit: Participants]
  [0, 6) Hours | 464 | 350 | 425 | 1239
  [6, 12) Hours | 114 | 104 | 106 | 324
  [12, 24) Hours | 84 | 72 | 86 | 242
  >=24 Hours | 43 | 45 | 30 | 118
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 339 | 292 | 316 | 947
  Male | 366 | 279 | 331 | 976

OUTCOME MEASURES:

1. Primary Outcome: Colonization at Day 1 Swab
Description: Was the swab collected on the day 1 visit (usually within 24 hours of birth) positive for any organism? If so, this is defined as positive.
Time Frame: First week of life
Population: Intention to Treat
Measure: Number; unit: Participants
Groups:
- CHX Cleansing - 7 Days: Babies in this group were born in clusters allocated to 7 days of chlorhexidine cleansing to the cord
- CHX Cleansing - 1 Day: Babies in this group were born in clusters allocated to 1 days of chlorhexidine cleansing to the cord
- Dry Cord Care: Babies in this group were born in clusters allocated to 0 days of chlorhexidine cleansing to the cord
Arm/Group | CHX Cleansing - 7 Days | CHX Cleansing - 1 Day | Dry Cord Care
Number analyzed (Participants) | 705 | 569 | 646
Participants
  Positive - one or more organisms found | 466 | 396 | 605
  Negative - no organisms found | 239 | 173 | 41
Statistical Analysis 1: Comparison: CHX Cleansing - 1 Day vs Dry Cord Care; Comparison of colonization prevalence, relative to dry cord care group; Test type: Superiority or Other; Binomial Regression, Log Link; General Estimating Equations (GEE) to account for clustered allocation; Prevalence Rate Ratio = 0.75, 95% CI 2-sided [0.70 to 0.81] — Prevalence Rate Ratio - Comparing Single CHX Cleansing to Dry Cord Care
Statistical Analysis 2: Comparison: CHX Cleansing - 7 Days vs Dry Cord Care; Comparison of colonization prevalence, relative to dry cord care group; Test type: Superiority or Other; Binomial Regression, Log Link; General Estimating Equations (GEE) to account for clustered allocation; Prevalence Rate Ratio = 0.71, 95% CI 2-sided [0.66 to 0.77] — Prevalence Rate Ratio - Comparing Multiple CHX Cleansing to Dry Cord Care

2. Primary Outcome: Colonization at Day 3 Swab
Description: Were any organisms found on the swab collected on at Day 03
Time Frame: First Week of Life
Population: Intent to Treat
Measure: Number; unit: Participants
Groups:
- CHX Cleansing - 7 Days: Babies in this group were born in clusters allocated to 7 days of chlorhexidine cleansing of the cord
- CHX Cleansing - 1 Day: Babies in this group were born in clusters allocated to 1 days of chlorhexidine cleansing of the cord
- Dry Cord Care: Babies in this group were born in clusters allocated to 0 days of chlorhexidine cleansing of the cord
Arm/Group | CHX Cleansing - 7 Days | CHX Cleansing - 1 Day | Dry Cord Care
Number analyzed (Participants) | 614 | 501 | 578
Participants
  Positive for any organisms | 363 | 381 | 563
  Negative for any organisms | 251 | 120 | 15
Statistical Analysis 1: Comparison: CHX Cleansing - 1 Day vs Dry Cord Care; Comparison of colonization prevalence, relative to dry cord care group; Test type: Superiority or Other; Binomial Regression, Log Link; Generalized Estimating Equations to account for clustered allocation; Prevalence Rate Ratio = 0.78, 95% CI 2-sided [0.74 to 0.82] — Prevalence Ratio Ratio - Comparing Single Cleansing to Dry Cord Care
Statistical Analysis 2: Comparison: CHX Cleansing - 7 Days vs Dry Cord Care; Comparison of colonization prevalence, relative to dry cord care group; Test type: Superiority or Other; Binomial Regression, Log Link; Generalized Estimating Equations to account for clustered allocation; Prevalence Rate Ratio = 0.61, 95% CI 2-sided [0.57 to 0.65] — Prevalence Rate Ratio - Comparing Multiple Cleansing to Dry Cord Care

3. Primary Outcome: Colonization at Day 7 Swab
Description: Were any organisms found on the swab collected on the day 07 visit?
Time Frame: First Week of Life
Population: Intent to Treat
Measure: Number; unit: Participants
Arm/Group | CHX Cleansing - 7 Days | CHX Cleansing - 1 Day | Dry Cord Care
Number analyzed (Participants) | 593 | 467 | 561
Participants
  Positive for any organisms | 328 | 415 | 540
  Negative for any organisms | 265 | 52 | 21
Statistical Analysis 1: Comparison: CHX Cleansing - 1 Day vs Dry Cord Care; Comparison of colonization prevalence, relative to dry cord care group; Test type: Superiority or Other; Binomial Regression, Log Link; General Estimating Equations to adjust for clustered allocation; Prevalence Rate Ratio = 0.92, 95% CI 2-sided [0.89 to 0.96] — Prevalence Rate Ratio - Comparing Single Cleansing to Dry Cord Care
Statistical Analysis 2: Comparison: CHX Cleansing - 7 Days vs Dry Cord Care; Comparison of colonization prevalence, relative to dry cord care group; Test type: Superiority or Other; Binomial Regression, Log Link; General Estimating Equations to account for clustered allocation; Prevalence Rate Ratio = 0.57, 95% CI 2-sided [0.53 to 0.63] — Prevalence Ratio Ratio - Comparing Multiple Cleansing to Dry Cord Care

ADVERSE EVENTS:
Arm/Group | CHX Cleansing - 7 Days | CHX Cleansing - 1 Day | Dry Cord Care
Serious Adverse Events (participants affected / at risk) | 0/705 | 0/571 | 0/647
Other Adverse Events (participants affected / at risk) | 0/705 | 0/571 | 0/647

LIMITATIONS AND CAVEATS:
Not all possible swab data were available for each baby due to staff leave/holiday, unplanned work stoppage, child/mother absent/moved/died, swab collected but not processed - these reasons did not differ between the groups

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No